CLINICAL TRIAL: NCT06553196
Title: MATAspire: Mental Health Awareness Tailored App for Substance Prevention and Integrated Resilience Education
Acronym: MATAspire
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: California State University, Northridge (Other)
Responsible Party: Principal Investigator, Bethany Rainisch, Principal Investigator, Department Chair, Professor, California State University, Northridge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H79SP083737
Record Dates: First submitted 2024-08-08; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Alcohol Use; Cannabis Use; Nicotine Use; Illicit Drug Use; Prescription Opioid Misuse
MeSH Terms: conditions — Alcohol Drinking; Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prevention group (Experimental): Web-app with 6 weekly coping & substance modules
  Interventions: Behavioral: MATAspire Web-app
- Control Group (No Intervention): No access to web-app

INTERVENTIONS:
Behavioral: MATAspire Web-app — Substance misuse prevention education and adaptive coping skills
  Arms: Prevention group

SUMMARY:
The MATAspire intervention is a web-app designed to promote substance misuse prevention education and bolster protective coping skills whereby students complete six weekly interactive modules using a smart device or computer. Each module is approximately 15-20 minutes long and focuses on select substances and coping strategies: (i) adaptive coping strategies, (ii) alcohol, (iii) cannabis, (iv) nicotine, (v) prescription drugs and opioids, (vi) final module. The modules are based on key theoretical constructs, behavior change strategies, and practical module components: attitudes (knowledge), perceived susceptibility (risk perceptions), and subjective norms (normative re-education). The intervention will be evaluated via a time series design using a sample of (~1000 students) randomly assigned to either the intervention or the control conditions at a public institution in Southern California.

ELIGIBILITY:
Inclusion Criteria:

* Current Cal State Northridge (CSUN) matriculated students with active CSUN email
* Age 18 and older

Exclusion Criteria:

* Not currently a CSUN student
* CSUN students under the age of 18 years
* Have previously participated in this study
* Identified as having an alcohol or substance use disorder (AUD or SUD) as determined by the brief Diagnostic and Statistical Manual of Mental Disorders (DSM) 5 screener

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2024-08-24 (Estimated); Primary Completion 2028-05-15 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline alcohol use behavior at 3 months | Baseline and 90-days following intervention completion
  Measured as the number of days drinking alcohol in past 30-days
Change from baseline binge drinking at 3 months | Baseline and 90-days following intervention completion
  Measured as the number of days consumed five or more alcoholic beverages at the same time for males; four or more for females in past 30-days
Change from baseline cannabis use at 3 months | Baseline and 90-days following intervention completion
  Measured as the number of days smoking, vaping, dabbing, oral (edibles/gummies/drinks), sprays, tinctures, and topically in past 30-days
Change from baseline nicotine use at 3 months | Baseline and 90-days following intervention completion
  Measured as the number of days using menthol cigarettes, regular cigarettes, loose tobacco rolled into cigarettes or cigars, pipe tobacco, snuff, chewing tobacco, dipping tobacco, snus, and others in past 30-days
Change from baseline electronic vape use products at 3 months | Baseline and 90-days following intervention
  Measured as the number of days using vaporizers, vape pens, hookah pens, electronic cigarettes, e-pens, or electronic nicotine delivery systems in past 30-days
Change from baseline non-prescribed prescription drug use behavior at 3 months | Baseline and 90-days following intervention completion
  Measured as the number of days used stimulants, sedatives, benzodiazepines, and prescription opioids in past 30-days
Change from baseline coping skills at 3 months | Baseline and 90-days following intervention completion
  Measured as the degree of effective and ineffective ways to cope with a stressful life event in ...

SECONDARY OUTCOMES:
Change from baseline alcohol use related outcomes at 3 months | Baseline and 90-days following intervention completion
  Measured as participants who report any past 30-day alcohol use indicate how many times they have experienced select outcomes in the last 30 days while drinking alcohol, or as a result of their alcohol use
Change from baseline nicotine use related outcomes at 3 months | Baseline and 90-days following intervention completion
  Measured as participants who report any past 30-day nicotine use indicate how many times they have experienced ten select outcomes in the last 30 days while using nicotine, or as a result of their nicotine use.
Change from baseline cannabis use related outcomes at 3 months | Baseline and 90-days following intervention completion
  Measured as participants who report any past 30-day cannabis use indicate how many times they have experienced ten select outcomes in the last 30 days while using cannabis, or as a result of their cannabis use
Change from baseline non-prescribed prescription drug use related outcomes at 3 months | Baseline and 90-days following completion of intervention
  Measured as participants who report any past 30-day non-prescribed prescription drug use indicate how many times they have experienced ten select outcomes in the last 30 days while using prescription drugs not prescribed to them, or for the purpose of feeling or experiencing something

OTHER OUTCOMES:
Change from baseline risk perceptions at 3 months | Baseline and 90-days following intervention completion
  Measured by participants' evaluation of their perceived risk level for the following substance use behaviors: nicotine use once or twice a week, binge drinking daily, binge drinking once or twice a week, cannabis or marijuana use once or twice a week, electronic vape products once or twice a week, opioid drugs once or twice a week, non-prescribed prescription drugs once or twice a week. Response options for each behavior include 1='no risk', 2='slight risk', 3='moderate risk', 4='great risk'.
Change from baseline subjective norms at 3 months | Baseline and 90-days following intervention completion
  Measured by participants' indication of what percentage of students on campus they perceive use a variety of substances within the last 30 days (i.e. alcohol, cannabis, tobacco or nicotine delivery products, prescription stimulants, sedatives or sleeping pills, prescription opioids, and hallucinogens) choosing one of ten percentile intervals from 0-100%.
Change from baseline attitudes at 3 months | Baseline and 90-days following intervention completion
  Measured by participants' attitude or feeling towards using mental health and substance use services on campus. Responses range from agree to disagree.
Physical Activity | Baseline and 90-days following intervention completion
  Measured by participants' indication of number of days of exercise in past week exercising. Examples of exercise are 'going to the gym', 'running', 'swimming', 'hiking', 'lifting weights or toning muscles', 'going for a brisk walk', or 'dancing', etc.
Sleep | Baseline and 90-days following intervention completion
  Measured as participants' report of average number of hours of sleep on a weeknight, excluding naps, over the past. Response options are 'less than 4 hours', '4 hours', '5 hours', '6 hours', '7 hours', '8 hours', '9 hours', '10 hours or more', or prefer not to answer.
Nutrition | Baseline and 90-days following intervention completion
  Measured as participants' report of past week average number of servings of fruit and average number of servings of vegetables consumed.
Socio-demographics | Baseline
  Participant characteristics, including age, Hispanic origin, race, sex at birth, gender identification, sexual orientation, living situation, college status, military service/veteran status, arrest history, parole/probation status, and household income
Adverse Childhood Experiences (ACE) | Baseline
  ACE are conceptualized as maltreatment (e.g., verbal, emotional, physical, and sexual abuse), and household dysfunction (e.g., parent/caregiver substance use, intimate partner violence, incarceration, homelessness, mental illness, separation/divorce. Participants respond to each of the ten ACE items as 1=Yes or 0=No. An ACE score will be computed with a range from 0-10.
Developmental Transition | Baseline
  Participants respond 1=Yes or 0=No to a list of 18 major life events within the last three years. Example life events include: getting into a new romantic relationship; breaking up with a girlfriend or boyfriend; losing a job; being unemployed and not able to find work; caring for a parent or relative; getting extremely ill; having a baby; losing a baby; or having family separated due to immigration. A total score will be computed with a range from 0-18.
Anxiety | Baseline and 90-days following intervention completion
  The Generalized Anxiety Disorder 7-item (GAD-7) is a screening tool for generalized anxiety disorder. This is calculated by assigning scores of 0, 1, 2, and 3 to the response categories below, respectively, of "not at all," "several days," "more than half the days," and "nearly every day." GAD-7 total score for the seven items ranges from 0 to 21. Higher scores indicate more anxiety.
  Participants' will indicate how often they felt they were/had 'nervous anxious or on edge', 'not able to stop or control worrying', 'worrying too much about different things', 'trouble relaxing', 'being so restless it was hard to sit still', 'become easily annoyed or irritable', over the past 2 weeks.
Depression | Baseline and 90-days following intervention completion
  The Center for Epidemiological Studies-Depression (CES-D)10-item scale assesses depressive symptoms in the past week. Participants will indicate how often (rarely=0, some/little=1, occasionally=2, most of the time=3) they felt 'bothered by things that usually don't bother me', 'they had trouble keeping their mind on what they were doing', 'depressed', 'everything was an effort', 'hopeful about the future', 'fearful', 'sleep was restless', 'happy', 'lonely', 'they could not get going' in last week.
  Items 5 and 8 are reverse coded. The total score is calculated by totaling all items scored after reversing the positive mood items. Possible range for scores is 0-30 with higher scores representing greater degrees of depressed mood.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Project website — https://www.csun.edu/mataspire